CLINICAL TRIAL: NCT05671133
Title: Effectiveness and Implementation of a Clinician Decision Support System to Prevent Suicidal Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthew K. Nock, PhD, Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022P002689
Record Dates: First submitted 2022-12-16; First posted 2023-01-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Suicide; Suicide, Attempted
MeSH Terms: conditions — Suicide; Suicide, Attempted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Patient's clinician is given Clinician Decision Support Tool
  Interventions: Diagnostic Test: Clinician Decision Support Tool
- Control (No Intervention): Patient's clinician is not given Clinician Decision Support Tool (care as usual)

INTERVENTIONS:
Diagnostic Test: Clinician Decision Support Tool — Clinician Decision Support Tool that provides information about patient's statistical probability of suicide attempt in next 1 month
  Arms: Experimental

SUMMARY:
The primary aim of this project are to evaluate a comprehensive, practice-ready, and deployment-focused strategy for improving the prediction and prevention of suicide attempts among a sample of 4,000 patients presenting to an ED with a psychiatric concern. Our first aim is to evaluate the effects of providing information about risk of patient suicidal behavior to ED clinicians. We hypothesize that patients randomly assigned to have their clinician receive their risk score will have a lower rate of suicide attempts during 6-month follow-up and that this effect will be mediated by changes in clinician decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presentation to emergency psychiatry service

Exclusion Criteria:

* Inability to understand study procedures and provide informed consent, such as those with gross cognitive impairment (including florid psychosis), intellectual disability, dementia, acute intoxication
* Presence of violent or extremely agitated behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Suicide attempt | 6-months
  Suicide attempts will be measured using two methods: (a) self-report surveys and (b) documentation in the Electronic Health Record during the follow-up period. Self-report questions about suicide attempts will be those from the Self-Injurious Thoughts and Behaviors Interview (SITBI), a widely-used measure of suicidal thoughts and behaviors with strong reliability and validity and one of the measures recommended in the PhenX toolkit. We also will examine all new medical records during the 6-months following each participant's index ED visit to determine if the participant revisited the hospital due to suicide ideation or suicide attempt during the follow-up period. This approach has been used in prior studies to measure such outcomes. In our own prior work in the ED we have found high agreement between self-reports on the SITBI and the documentation of suicide attempts in electronic medical records (K=.84).

SECONDARY OUTCOMES:
Suicide attempt | 1-month
  Secondary endpoints are suicide attempt (using the same assessment methods as the primary endpoint) within 1-month post-randomization and will also be assessed using two sample tests of proportions.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared via the National Institute of Mental Health National Data Archive
Supporting Information: Study Protocol, SAP
Time Frame: By study end